CLINICAL TRIAL: NCT06248463
Title: Automatic Blood Pressure Assessment in Waiting Room During Pregnancy Compare to 24-h Ambulatory Blood Pressure Measurement
Brief Title: Blood Pressure Assessment in Waiting Room During Pregnancy
Acronym: WAPA-Pregnan
Status: Not yet recruiting | Type: Observational
Sponsor: Fundación para la Formación e Investigación de los Profesionales de la Salud de Extremadura (Other)
Collaborators: University of Salamanca (Other)
Responsible Party: Sponsor
Other Study IDs: FUNDESALUD
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-01

CONDITIONS: Hypertension; Pregnancy Induced Hypertension
Keywords: Hypertension in pregnancy.; Blood Pressure measurement.
MeSH Terms: conditions — Hypertension; Hypertension, Pregnancy-Induced

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Woman with hypertension risk related to gestation: SBP readings above 130 mmHg in office or the presence of a risk factor for eclampsia: (hypertensive disease in previous pregnancy, chronic hypertension, chronic renal disease, diabetes mellitus, or autoimmune disease) or any two moderate-risk factors (nulliparity, age ≥40 years, BMI ≥35 kg/m2, family history of PE, or interpregnancy interval >10 years)
  Interventions: Diagnostic Test: BP measurement in waiting room for 20 minutes

INTERVENTIONS:
Diagnostic Test: BP measurement in waiting room for 20 minutes — Measured of BP will be performance in waiting room for 20 minutes every 3 minutes and report by an mobile app. After 24h-ABPM device will be implanted. Results of SBP and DBP obtained in office will be compared with 24-h, diurnal and nocturnal SBP/DBP mean.
  BP will be measured automatically and repeatedly every 3 minutes in the waiting room for 20 minutes. Subsequently, a SpaceLab ABPM monitor will be implanted.
  Other Names: ABPM-24 h

SUMMARY:
The goal of this observational study is to compare in healthy pregnant women during the first trimester. The main question it aims to answer are:

Accuracy of measuring automatically Blood Pressure (BP) at appointment compared to 24 Hour Ambulatory Blood Pressure Monitor (ABPM).

Participants will be BP measured with homologated device every 3 minutes in waiting room for 20 minutes.

Researchers will compare Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) in clinical visit to see if are comparable to ABPM.

DETAILED DESCRIPTION:
659 pregnant women will be recruitment if they In with SBP readings above 130 mmHg in office or the presence of a risk factor for eclampsia: (hypertensive disease in previous pregnancy, chronic hypertension, chronic renal disease, diabetes mellitus, or autoimmune disease) or any two moderate-risk factors (nulliparity, age ≥40 years, BMI ≥35 kg/m2, family history of PE, or interpregnancy interval >10 years).

Measured of BP will be performance in waiting room for 20 minutes every 3 minutes and report by an mobile app. After 24h-ABPM device will be implanted. Results of SBP and DBP obtained in office will be compared with 24-h, diurnal and nocturnal SBP/DBP mean.

BP will be measured automatically and repeatedly every 3 minutes in the waiting room for 20 minutes. Subsequently, a SpaceLab ABPM monitor will be implanted. The SBP and DBP results obtained in the waiting room will be compared with the ABPM results.

Clinical data related to eclampsia and maternal and newborn pregnancy outcomes will be collected from all patients.

ELIGIBILITY:
Inclusion Criteria:

Woman during the first 12 weeks of pregnancy Maternal age>35 Nulliparity Previous history of hypertension Short and long interpregnancy interval Use of assisted reproductive technologies Family history of preeclampsia Obesity. BMI>30. Hyperglycemia Renal disease

Exclusion Criteria:

Any inability to perform 24-h ambulatory BP measurement

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Gestation
Study Population: Pregnant women with suspected hypertension
Sampling Method: Non-Probability Sample
Enrollment: 659 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Differences in Blood Pressure between office and 24- Ambulatory Blood Pressure Meassurement (24-h ABPM) | 10 mounths
  Concordance of Systolic and Diastolic Blood Pressure mean between waiting room and 24-h ABMP measurements
Maternal | 10 months
  Cardiovascular events, preeclampsia, abruptio, cesarean delivery, hemorrhage,pulmonary edema, death
Newborn | 10 monts
  Growth restriction, preterm delivery, congenital anomalies, stillbirth, neonatal death.